CLINICAL TRIAL: NCT03113695
Title: Obinutuzumab, High Dose Methylprednisolone (HDMP), and Lenalidomide for the Treatment of Patients With Richter's Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Thomas Kipps, Deputy Director, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161265
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Richter's Syndrome; CLL
Keywords: Richter's Syndrome; CLL; Chronic Lumphocytic Leukemia; obinutuzumab; HDMP; lenalidomide; cancer; methylprednisolone
MeSH Terms: conditions — Neoplasms | interventions — obinutuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- obinutuzumab, lenalidomide, and HDMP (Experimental)
  Interventions: Drug: Obinutuzumab; Drug: lenalidomide; Drug: HDMP

INTERVENTIONS:
Drug: Obinutuzumab — obinutuzumab 1000 mg x 8 doses (first dose split on Cycle 1 days 1 100mg and 2 900mg; then day 8 and 15 of cycle 1; then day 1 of cycles 2-6, each cycle being 28 days long)
Drug: lenalidomide — lenalidomide PO daily. The starting dose of lenalidomide is 5 mg PO daily. Starting on C2D1, the dose increases every 2 weeks in 5 mg increments to a maximum of 25 mg PO daily. Patients will continue lenalidomide until disease progression, unacceptable toxicity, or subsequent therapy.
Drug: HDMP — methylprednisolone 1000 mg/m2 (ie HDMP) on days 1-5 of cycles 1-4

SUMMARY:
The purpose of the study is to investigate whether combination of obinutuzumab, lenalidomide, and high dose methylprednisolone in the treatment of Richter's Syndrome. The study will evaluate whether this regimen can reduce the amount of cancerous cells in your body. All of these agents are approved by the FDA Obinutuzumab is a protein molecule manufactured from a single cell population, has been approved by the Food and Drug Administration (FDA) for the treatment of CLL of SLL. Lenalidomide is for the treatment of patients with other blood cancers. Methylprednisolone is a type of steroid, and it is used in a wide variety of medical conditions. These agents and the combination of these agents are not approved for the treatment of Richter's Syndrome and are considered experimental.

DETAILED DESCRIPTION:
This is a phase I trial to determine the safety and tolerability of the combination of obinutuzumab, lenalidomide, and HDMP for patients with RS. There is not a standard of care for patients with Richter's Syndrome (RS). Ten patients will be enrolled with RS diagnosed by histology or flow cytometry and CLL, regardless of prior treatment for either condition.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of Richter's Syndrome (RS)
* No requirement nor restriction for prior therapy or stage
* Measurable disease: may include FDG avid lesion, lymph node greater than 1.5 cm in greatest diameter, or clonal large B-cells in peripheral blood or bone marrow.
* ECOG 0-2
* Adequate organ function
* Adequate bone marrow function

Lenalidomide-related inclusion criteria:

* Able to take aspirin (81mg or 325mg) daily, warfarin, low molecular weight heparin, or equivalent anticoagulation as prophylactic medication.
* All study participants must be registered into the mandatory REVLIMID REMS® program, and be willing and able to comply with the requirements of REMS®.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 10 - 14 days prior to and again within 24 hours prior to starting REVLIMID® and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking REVLIMID®. FCBP must also agree to ongoing pregnancy testing.
* Males must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known hypersensitivity to any of the study drugs
* Patients with a malignancy that has been treated, but not with curative intent, will be excluded, unless the malignancy has been in remission without treatment for 2 years prior to enrollment.
* Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks before the start of treatment
* Major surgery within 4 weeks prior to the start of treatment
* Known infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus 1 (HTLV-1) seropositive status
* Positive hepatitis serology
* Women who are pregnant or lactating
* Vaccination with a live vaccine a minimum of 28 days prior to the start of treatment
* Uncontrolled diabetes mellitus
* Myocardial infarction within 6 months of starting study drug
* Other clinically significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the combination of obinutuzumab, lenalidomide, and high dose methylprednisolone in treatments with Richter's Syndrome (RS) measured Via Adverse Events | 2 years
  Measured Via Adverse Events

SECONDARY OUTCOMES:
Overall response rate of RS and CLL | 12 months and 24 months
  Measure via the Cheson Criteria for response in lymphoma.
Progression-free survival rate | 12 months and 24 months
  Measure via the Cheson Criteria for response in lymphoma. PFS is defined as the time from entry onto a study until lymphoma progression or death as a result of any cause.
Overall survival rate | 12 months and 24 months
  Measure via the Cheson Criteria for response in lymphoma. Defined as the time from entry onto the clinical trial until death as a result of any cause.
Patients able to receive a subsequent stem cell transplant (percentage) | 12 months and 24 months
  Measure by percentage of patients able to receive subsequent tell cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Kipps, M.D., Ph.D., Principal Investigator — University of California
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No